CLINICAL TRIAL: NCT00651664
Title: A Phase I Clinical and Pharmacodynamic Study of MLN8237, A Novel Aurora A Kinase Inhibitor, in Patients With Advanced Malignancies
Brief Title: A Phase I Clinical and Pharmacodynamic Study of MLN8237, A Novel Aurora A Kinase Inhibitor, in Participants With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C14002; 2006-006048-68 (EudraCT Number); U1111-1187-1151 (Registry Identifier: WHO)
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-11

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Alisertib 5 mg QD 7D (Experimental): Alisertib 5 mg, capsules, orally, once daily (QD) for 7 days (D) followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 3 cycles).
  Interventions: Drug: alisertib
- Alisertib 80 mg QD 7D (Experimental): Alisertib 80 mg, capsules, orally, QD for 7 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 4 cycles).
  Interventions: Drug: alisertib
- Alisertib 150 mg QD 7D (Experimental): Alisertib 150 mg, capsules, orally, QD for 7 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles).
  Interventions: Drug: alisertib
- Alisertib 50 mg BID 7D (Experimental): Alisertib 50 mg, capsules, orally, twice daily (BID) for 7 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 29 cycles).
  Interventions: Drug: alisertib
- Alisertib 60 mg BID 7D (Experimental): Alisertib 60 mg, capsules, orally, BID for 7 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles).
  Interventions: Drug: alisertib
- Alisertib 75 mg BID 7D (Experimental): Alisertib 75 mg, capsules, orally, BID for 7 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 8 cycles).
  Interventions: Drug: alisertib
- Alisertib 100 mg BID 7D (Experimental): Alisertib 100 mg, capsules, orally, BID for 7 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 21 cycles).
  Interventions: Drug: alisertib
- Alisertib 50 mg QD 14D (Experimental): Alisertib 50 mg, capsules, orally, QD for 14 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 25 cycles).
  Interventions: Drug: alisertib
- Alisertib 50 mg QD 21D (Experimental): Alisertib 50 mg, capsules, orally, QD for 21 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 10 cycles).
  Interventions: Drug: alisertib
- Alisertib 70 mg QD 21D (Experimental): Alisertib 70 mg, capsules, orally, QD for 21 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 2 cycles).
  Interventions: Drug: alisertib

INTERVENTIONS:
Drug: alisertib — Alisertib (MLN8237) capsules
  Other Names: MLN8237

SUMMARY:
This is a multicenter, dose escalation, phase 1 study of MLN8237 in adult participants with advanced malignancies (excluding those with primary bone marrow involvement, such as leukemias and multiple myeloma).

DETAILED DESCRIPTION:
The drug tested in this study is called alisertib. Alisertib is being tested to treat people who have advanced malignancies. This study determined the dose-limiting toxicity, maximum tolerated dose, safety and pharmacokinetics (how the drug moves through the body) for alisertib when given once or twice a day for 7 to 21 days.

This open label study enrolled 59 patients. Participants were enrolled in one of 10 dose escalation arms:

* Alisertib 5 mg once daily (QD) for 7 Days (D)
* Alisertib 80 mg QD 7D
* Alisertib 150 mg QD 7D
* Alisertib 50 mg twice daily (BID) 7D
* Alisertib 60 mg BID 7D
* Alisertib 75 mg BID 7D
* Alisertib 100 mg BID 7D
* Alisertib 50 mg QD 14D
* Alisertib 50 mg QD 21D
* Alisertib 70 mg QD 21D

All participants received treatment until their disease progressed or they experienced unacceptable alisertib-related toxicity.

This multi-center trial was conducted in Spain. The overall time to participate in this study was 730 days. Participants made multiple visits to the clinic, including a final visit 30 days after receiving their last dose of alisertib for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed metastatic and/or advanced malignancy (including lymphomas but excluding malignancies with extensive bone marrow involvement such as leukemias and multiple myeloma) for which standard treatment does not offer curative or life-prolonging potential.
2. Aged 18 years or more.
3. Eastern Cooperative Oncology Group performance status 0 or 1.
4. Have an expected survival longer than 3 months from enrollment in the study.
5. Radiographically or clinically evaluable tumor.
6. Suitable venous access for the conduct of blood sampling.
7. Recovered from the reversible effects of prior antineoplastic therapy (with the exception of alopecia and grade 1 neuropathy) with at least 4 weeks elapsed since the last exposure to cytotoxic chemotherapy or to radiotherapy and at least 6 weeks elapsed since exposure to nitrosoureas or mitomycin C. Participants treated with fully human monoclonal antibodies must not have received treatment with such antibodies for at least 6 weeks, and those treated with chimeric monoclonal antibodies must not have received treatment with such antibodies for at least 4 weeks. Participants treated with noncytotoxic small molecule drugs (eg, tyrosine kinase inhibitors, such as Tarceva® [erlotinib], and hormonal agents, such as Femara® [letrozole]) must not have received treatment with these drugs for at least 2 weeks before the first dose of alisertib was given.
8. Male participants must use an appropriate method of barrier contraception and inform any sexual partners that they must also use a reliable method of contraception from the time of informed consent until 3 months after the last dose of study treatment.
9. Female participants must be postmenopausal at least 1 year, OR surgically sterile, OR if of childbearing potential, agree to 2 effective methods of nonhormonal contraception, or agree to completely abstain from heterosexual intercourse.
10. Able to give written consent.

Exclusion Criteria:

1. Pregnant or lactating.
2. Major surgery or serious infection within the 28 days preceding the first dose of study treatment.
3. Life-threatening or uncontrolled medical illness unrelated to cancer.
4. Ongoing nausea or vomiting of any severity.
5. >Grade 1 diarrhea. Participants who require ongoing therapy with an antimotility agent to control diarrhea to a Grade 1 or lower level are not allowed to participate in this trial.
6. Known gastrointestinal disease or gastrointestinal procedures that could interfere with the oral absorption or tolerance of MLN8237.
7. History of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness such as severe chronic obstructive pulmonary disease.
8. Difficulty swallowing capsules.
9. Inability to take nothing by mouth except for water and prescribed medications for 2 hours before and 1 hour after each dose of MLN8237.
10. Received more than 4 previous cytotoxic chemotherapeutic regimens, including regimens used as adjuvant or neo-adjuvant therapies (in participants with metastatic breast cancer, a total of 5 previous cytotoxic chemotherapeutic regimens is permitted).
11. Prior treatment with high-dose chemotherapy, defined as chemotherapy requiring the use of peripheral blood or bone marrow stem cell support for hematopoietic reconstitution.
12. Prior treatment with radiation therapy involving ≥25% of the hematopoietically active bone marrow for the distribution of active bone marrow in adults).
13. Clinical and/or radiographic evidence of cerebral metastases. However, participants who have a history of central nervous system metastasis but who have no radiographic or clinical evidence of residual tumor (eg, following complete surgical resection or stereotactic radiosurgery) are not excluded from participation in this study.
14. Absolute neutrophil count(ANC) < 1500/mm^3; platelet count< 100,000/mm^3.
15. Serum creatinine >1.6 mg/dL or a measured or estimated (Cockcroft-Gault formula) creatinine clearance <40 mL/min
16. Bilirubin >1.5 times the upper limit of the normal range (ULN); aspartate aminotransferase(AST)/alanine aminotransferase(ALT) >2.5 times the ULN, and alkaline phosphatase(ALP) >2.5 times the ULN. Both the AST and ALP could be elevated up to 5 times the ULN if their elevation could be reasonably ascribed to the presence of metastatic disease to liver and/or to bone; however, the ALT in all circumstances must have been <2.5 times the ULN.
17. Abnormalities on 12-lead electrocardiogram considered by the investigator to be clinically significant or baseline prolongation of the rate-corrected QT interval (eg, repeated demonstration of QTc interval >450 milliseconds).
18. Known history of human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C.
19. Less than 4 weeks between the last dose of an investigational agent and the first dose of MLN8237.
20. Admission or evidence of benzodiazepine dependence or abuse and/or alcohol abuse or an inability to restrict consumption of alcohol to no more than 1 standard unit of alcohol per day during the study and for 30 days from the last dose of study treatment.
21. Activated partial thromboplastin time (aPTT) and/or prothrombin time (PT) exceeding the upper limit of the normal range.
22. Known bleeding diathesis or history of abnormal bleeding.
23. Ongoing therapy with an anticoagulant (e.g., aspirin, plavix, coumadin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-10-22 (Actual); Primary Completion 2010-09-01 (Actual); Study Completion 2011-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (2):
- Spain (2):
  - Ciutat Sanitaria Vall d'Hebron - Servicio de Oncologia, Barcelona
  - H. Clínico Universitario de Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Spain from 22 October 2007 to 05 April 2011.
Pre-assignment Details: Participants with a diagnosis of advanced malignancies were enrolled in a dose escalation study, alisertib 5, 80 150 mg once daily (QD) for 7 days; 50, 60, 75, 100 mg twice daily for 7 days; 50 mg QD for 14 days; 50, 70 mg QD for 21 days.
Groups:
- Alisertib 5 mg QD 7D: Alisertib 5 mg, capsules, orally, once daily (QD) for 7 days (D) followed by a 14-day recovery period in each 21-day cycle until disease progression or unacceptable alisertib-related toxicity (up to 3 cycles).
- Alisertib 80 mg QD 7D: Alisertib 80 mg, capsules, orally, QD for 7 days followed by a 14-day recovery period in each 21-day cycle until disease progression or unacceptable alisertib-related toxicity (up to 4 cycles).
- Alisertib 150 mg QD 7D: Alisertib 150 mg, capsules, orally, QD for 7 days followed by a 14-day recovery period in each 21-day cycle until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles).
- Alisertib 50 mg BID 7D: Alisertib 50 mg, capsules, orally, twice daily (BID) for 7 days followed by a 14-day recovery period in each 21-day cycle until disease progression or unacceptable alisertib-related toxicity (up to 29 cycles).
- Alisertib 60 mg BID 7D: Alisertib 60 mg, capsules, orally, BID for 7 days followed by a 14-day recovery period in each 21-day cycle until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles).
- Alisertib 75 mg BID 7D: Alisertib 75 mg, capsules, orally, BID for 7 days followed by a 14-day recovery period in each 21-day cycle until disease progression or unacceptable alisertib-related toxicity (up to 8 cycles).
- Alisertib 100 mg BID 7D: Alisertib 100 mg, capsules, orally, BID for 7 days followed by a 14-day recovery period in each 21-day cycle until disease progression or unacceptable alisertib-related toxicity (up to 21 cycles).
- Alisertib 50 mg QD 14D: Alisertib 50 mg, capsules, orally, QD for 14 days followed by a 14-day recovery period in each 28-day cycle until disease progression or unacceptable alisertib-related toxicity (up to 25 cycles).
- Alisertib 50 mg QD 21D: Alisertib 50 mg, capsules, orally, QD for 21 days followed by a 14-day recovery period in each 35-day cycle until disease progression or unacceptable alisertib-related toxicity (up to 10 cycles).
- Alisertib 70 mg QD 21D: Alisertib 70 mg, capsules, orally, QD for 21 days followed by a 14-day recovery period in each 35-day cycle until disease progression or unacceptable alisertib-related toxicity (up to 2 cycles).
Period: Overall Study
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D | Alisertib 50 mg QD 14D | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Started | 3 | 3 | 3 | 14 | 6 | 3 | 6 | 7 | 7 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 14 | 6 | 3 | 6 | 7 | 7 | 7
Not completed — Occurrence of Adverse Event(s) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Unsatisfactory Therapeutic Response | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Not completed — Progressive Disease | 3 | 3 | 3 | 12 | 4 | 1 | 3 | 6 | 5 | 5
Not completed — Patient Declined Further Treatment | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Reason not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all participants who received any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D | Alisertib 50 mg QD 14D | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D | Total
Number analyzed (Participants) | 3 | 3 | 3 | 14 | 6 | 3 | 6 | 7 | 7 | 7 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (9.07) | 62.3 (13.80) | 55.7 (20.79) | 62.5 (11.67) | 59.2 (18.74) | 48.3 (14.84) | 58.7 (8.69) | 58.0 (13.83) | 53.0 (11.08) | 64.7 (5.53) | 58.8 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 6 | 4 | 0 | 2 | 2 | 3 | 2 | 22
  Male | 3 | 2 | 1 | 8 | 2 | 3 | 4 | 5 | 4 | 5 | 37
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 3 | 3 | 3 | 14 | 6 | 3 | 6 | 7 | 6 | 5 | 56
  Not Hispanic/Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Race/Ethnicity, Customized [Number; unit: participants] — White
  participants | 3 | 3 | 3 | 14 | 6 | 3 | 6 | 7 | 7 | 7 | 59
Region of Enrollment [Number; unit: participants]
  Spain | 3 | 3 | 3 | 14 | 6 | 3 | 6 | 7 | 7 | 7 | 59
Height [Mean (Standard Deviation); unit: cm] | 164.0 (7.21) | 164.3 (10.79) | 167.3 (1.53) | 165.8 (9.26) | 160.5 (4.76) | 171.3 (10.26) | 165.2 (10.21) | 169.9 (10.92) | 160.4 (11.57) | 167.6 (8.40) | 165.4 (9.15)
Weight [Mean (Standard Deviation); unit: kg] | 83.7 (32.13) | 75.2 (10.56) | 70.3 (4.24) | 74.4 (16.48) | 64.8 (6.83) | 90.5 (7.74) | 69.6 (16.22) | 76.7 (15.06) | 69.1 (14.78) | 77.9 (11.91) | 74.0 (14.95)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — BSA = square root [ height (cm) x weight (kg) / 3600 ]
  m^2 | 1.93 (0.393) | 1.85 (0.191) | 1.81 (0.047) | 1.85 (0.225) | 1.70 (0.102) | 2.07 (0.098) | 1.78 (0.244) | 1.87 (0.204) | 1.75 (0.231) | 1.90 (0.145) | 1.84 (0.208)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT)
Description: DLT was evaluated using the National Cancer Institutes Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0; defined as any of the following events related to alisertib therapy:
  1. Grade 4 neutropenia lasting for ≥7 consecutive days during recovery
  2. Grade 4 neutropenia with fever and/or infection
  3. Confirmed platelet count <25,000/mm^3
  4. ≥Grade 3 nausea and/or emesis despite the use of an antiemetic prophylaxis
  5. ≥Grade 3 diarrhea that occurred despite therapy with loperamide
  6. Any other Grade 3 or greater nonhematologic toxicity, with the following exceptions: Grade 3 arthralgia/myalgias, Any grade of alopecia, Brief (< 1 week) Grade 3 fatigue
  7. Treatment delay of >1 week because of a failure of adequate hematologic or nonhematologic recovery from the previous cycle of treatment.
  8. Other alisertib-related nonhematologic toxicities ≥ Grade 2 that, in the opinion of the investigator, required a dose reduction or discontinuation of therapy with alisertib.
Time Frame: First dose through 30 days following the last dose of study drug (up to 730 days)
Population: DLT Evaluable Population was defined as all participants who received at least 75% of their planned alisertib doses for their first cycle of treatment (unless interrupted by DLT) and had sufficient follow-up data to allow the investigators and sponsor to determine whether DLT occurred.
Measure: Number; unit: participants
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D | Alisertib 50 mg QD 14D | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 6 | 2 | 6 | 6 | 7 | 6
participants | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 1 | 1 | 3

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Alisertib
Description: The MTD was defined as the highest dose at which DLT occurred in 0/3 or 1/6 participants.
Time Frame: Signing of the Informed Consent through 30 days following the last dose of study drug (up to 730 days)
Population: as for outcome 1
Measure: Number; unit: mg BID for 7 Days
Groups:
- Alisertib: Alisertib 5, 80 or 150 mg, capsules, orally, once daily (QD) for 7 days, followed by a 14-day recovery period or alisertib 50, 60, 75 or 100 mg, capsules, orally, twice daily (BID) for 7 days, followed by a 14-day recovery period or alisertib 50 mg, capsules, orally, QD for 14 days followed by a 14-day recovery period or alisertib 50 or 70 mg, capsules, orally, QD for 21 days followed by a 14-day recovery period in each cycle until disease progression or unacceptable alisertib-related toxicity (up to 29 cycles).
Arm/Group | Alisertib
Number analyzed (Participants) | 54
mg BID for 7 Days | 50

3. Secondary Outcome: Cmax: Maximum Observed Concentration for Alisertib 7 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 24 hour) post-dose on Day 1 and Pre-dose and multiple time-points (up to 10 hours) on Day 7
Population: Pharmacokinetic (PK) Evaluable Population was defined as all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis. Here number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar (nM)
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D
Number analyzed (Participants) | 3 | 3 | 3 | 14 | 6 | 3 | 6
nanomolar (nM)
  Day 1 | 123.15 (6.554) | 1774.12 (36.496) | 2014.81 (22.038) | 1035.3 (75.70) | 1536.1 (44.70) | 1266.6 (45.69) | 3196.4 (51.11)
  Day 7: number analyzed (Participants) | 3 | 3 | 3 | 10 | 6 | 3 | 5
  Day 7 | 109.13 (34.458) | 1502.89 (32.818) | 4136.24 (26.253) | 1964.4 (46.26) | 3412.5 (27.06) | 5710.4 (23.89) | 4694.2 (38.86)

4. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib 7 Day Dosing
Time Frame: as for outcome 3
Population: PK Evaluable Population was defined as all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis. Here number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Median (Full Range); unit: hour(hr)
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D
Number analyzed (Participants) | 3 | 3 | 3 | 14 | 6 | 3 | 6
hour(hr)
  Day 1 | 1.920 [1.58 to 2.00] | 2.730 [1.70 to 4.00] | 4.000 [2.00 to 5.90] | 2.040 [2.00 to 6.17] | 2.000 [2.00 to 4.08] | 2.000 [2.00 to 2.10] | 3.835 [1.98 to 4.08]
  Day 7: number analyzed (Participants) | 3 | 3 | 3 | 12 | 6 | 3 | 5
  Day 7 | 1.670 [1.00 to 1.97] | 1.580 [1.50 to 6.00] | 1.550 [1.42 to 3.43] | 2.000 [1.25 to 8.00] | 2.000 [0.92 to 4.00] | 4.170 [1.75 to 5.83] | 1.580 [1.00 to 6.00]

5. Secondary Outcome: AUCt: Area Under the Concentration-time Curve From Time 0 to Time t for Alisertib 7 Day Dosing
Time Frame: Cycle1: Pre-dose and multiple time-points (up to 24 hour) post-dose on Day 1 and Pre-dose and multiple time-points (up to 10 hours) on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hour(h)
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D
Number analyzed (Participants) | 3 | 3 | 3 | 14 | 6 | 3 | 6
nM*hour(h)
  Day 1: number analyzed (Participants) | 1 | 3 | 3 | 12 | 4 | 2 | 4
  Day 1 | 975.0 (NA) — CV was not calculated for 1 participant. | 18204.2 (36.19) | 27262.7 (38.0) | 6314.1 (82.32) | 9771.5 (53.77) | 6895.3 (9.21) | 16541.5 (65.99)
  Day 7: number analyzed (Participants) | 2 | 3 | 3 | 9 | 6 | 3 | 5
  Day 7 | 658.5 (35.64) | 16101.6 (38.81) | 48421.8 (36.53) | 17795.6 (43.87) | 25853.3 (41.44) | 51684.4 (24.87) | 40166.7 (51.90)

6. Secondary Outcome: Terminal Half-Life (t1/2) for Alisertib 7 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Day 7 or 8 (BID arms)
Population: Participants from the PK Evaluable Population, all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis. sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis, with data available for t1/2 analysis.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D
Number analyzed (Participants) | 0 | 2 | 3 | 9 | 6 | 3 | 6
hr |  | 18.25 (8.697) | 19.80 (6.129) | 15.913 (6.4766) | 19.475 (15.5019) | 18.500 (7.6295) | 13.637 (6.8712)

7. Secondary Outcome: Accumulation Ratio (Rac) for Alisertib 7 Day Dosing
Description: Rac for Day 7=AUCt Day 7/AUCt Day 1.
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Day 7
Population: Participants from the PK Evaluable Population, all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis, with data available for analysis Rac.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D
Number analyzed (Participants) | 1 | 3 | 3 | 8 | 4 | 2 | 4
ratio | 0.874 (0) | 0.892 (0.1331) | 1.954 (0.9092) | 2.295 (0.9846) | 2.583 (0.8959) | 7.765 (1.9163) | 2.350 (1.4926)

8. Secondary Outcome: Peak/Trough Ratio for Aliserib 7 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Day 7
Population: Participants from the PK Evaluable Population, all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis, with data available for analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D
Number analyzed (Participants) | 2 | 3 | 3 | 9 | 6 | 3 | 5
ratio | 5.950 (0.3253) | 4.650 (0.2163) | 4.507 (0.3029) | 3.083 (2.2296) | 3.050 (1.4056) | 1.867 (0.6009) | 2.256 (1.2013)

9. Secondary Outcome: CLss/F: Apparent Oral Clearance at Steady State 7 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Day 7
Population: Participants from the PK Evaluable Population, all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis, with data available for CLss/F analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter(L)/hr
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D
Number analyzed (Participants) | 3 | 3 | 3 | 9 | 6 | 3 | 5
liter(L)/hr | 14.055 (27.6995) | 9.604 (35.5110) | 5.967 (31.2592) | 5.414 (57.9221) | 4.182 (51.2761) | 2.795 (23.5794) | 4.798 (49.4182)

10. Secondary Outcome: Cmax: Maximum Observed Concentration for Alisertib 14 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 24 hour) post-dose on Day 1 and Pre-dose and multiple time-points (up to 10 hours) on Days 7 and 14
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 50 mg QD 14D
Number analyzed (Participants) | 7
nM
  Day 1 | 1145.4 (53.09)
  Day 7: number analyzed (Participants) | 6
  Day 7 | 1418.1 (70.96)
  Day 14: number analyzed (Participants) | 6
  Day 14 | 1671.1 (51.66)

11. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib 14 Day Dosing
Time Frame: as for outcome 10
Population: as for outcome 4
Measure: Median (Full Range); unit: hr
Arm/Group | Alisertib 50 mg QD 14D
Number analyzed (Participants) | 7
hr
  Day 1 | 2.030 [1.00 to 6.00]
  Day 7: number analyzed (Participants) | 6
  Day 7 | 2.000 [2.00 to 4.00]
  Day 14: number analyzed (Participants) | 6
  Day 14 | 2.000 [1.02 to 4.00]

12. Secondary Outcome: AUCt: Area Under the Concentration-time Curve From Time 0 to Time t for Alisertib 14 Day Dosing
Time Frame: as for outcome 10
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Alisertib 50 mg QD 14D
Number analyzed (Participants) | 7
nM*hr
  Day 1: number analyzed (Participants) | 5
  Day 1 | 15363.0 (24.82)
  Day 7: number analyzed (Participants) | 6
  Day 7 | 17918.8 (78.55)
  Day 14: number analyzed (Participants) | 6
  Day 14 | 16449.8 (59.87)

13. Secondary Outcome: Terminal Half-Life (t1/2) for Alisertib 14 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Days 7 and 14
Population: Participants from the PK Evaluable Population, all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis, with data for analysis of t1/2. No data was available for analysis at Day 7.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Alisertib 50 mg QD 14D
Number analyzed (Participants) | 5
hr | 26.62 (13.611)

14. Secondary Outcome: Accumulation Ratio (Rac) for Alisertib 14 Day Dosing
Description: Rac for Day 7=AUCt Day 7/AUCt Day 1. Rac for Day 14=AUCt Day 7/AUCt Day 1.
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Days 7 and 14
Population: Participants from the PK Evaluable Population, all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis, with data available for analysis Rac. Here number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 50 mg QD 14D
Number analyzed (Participants) | 7
ratio
  Day 7: number analyzed (Participants) | 5
  Day 7 | 1.671 (0.8242)
  Day 14: number analyzed (Participants) | 4
  Day 14 | 1.813 (0.5001)

15. Secondary Outcome: Peak/Trough Ratio for Aliserib 14 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Days 7 and 14
Population: Participants from the PK Evaluable Population, all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis, with data available for analysis. Here number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 50 mg QD 14D
Number analyzed (Participants) | 7
ratio
  Day 7: number analyzed (Participants) | 6
  Day 7 | 4.415 (2.5016)
  Day 14: number analyzed (Participants) | 6
  Day 14 | 7.412 (4.2472)

16. Secondary Outcome: CLss/F: Apparent Oral Clearance at Steady State 14 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Days 7 and 14
Population: Participants from the PK Evaluable Population, all participants for whom there were sufficient dosing and alisertib concentration-time data to permit noncompartmental PK analysis, with data available for CLss/F analysis. Here number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Alisertib 50 mg QD 14D
Number analyzed (Participants) | 7
L/hr
  Day 7: number analyzed (Participants) | 6
  Day 7 | 5.381 (92.8272)
  Day 14: number analyzed (Participants) | 6
  Day 14 | 5.856 (98.2758)

17. Secondary Outcome: Cmax: Maximum Observed Concentration for Alisertib 21 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 24 hour) post-dose on Day 1 and Pre-dose and multiple time-points (up to 10 hours) on Days 14 and 21
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Number analyzed (Participants) | 7 | 7
nM
  Day 1 | 1112.3 (42.99) | 2220.3 (47.57)
  Day 14: number analyzed (Participants) | 7 | 5
  Day 14 | 1524.1 (64.25) | 2595.0 (42.98)
  Day 21: number analyzed (Participants) | 6 | 4
  Day 21 | 1651.7 (30.70) | 2093.7 (11.68)

18. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib 21 Day Dosing
Time Frame: as for outcome 17
Population: as for outcome 4
Measure: Median (Full Range); unit: hr
Arm/Group | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Number analyzed (Participants) | 7 | 7
hr
  Day 1 | 4.000 [2.00 to 6.17] | 2.000 [2.00 to 2.02]
  Day 14: number analyzed (Participants) | 7 | 5
  Day 14 | 2.070 [1.00 to 4.00] | 2.130 [2.00 to 5.08]
  Day 21: number analyzed (Participants) | 6 | 4
  Day 21 | 2.100 [2.00 to 24.80] | 2.125 [2.00 to 2.33]

19. Secondary Outcome: AUCt: Area Under the Concentration-time Curve From Time 0 to Time t for Alisertib 21 Day Dosing
Time Frame: as for outcome 17
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Number analyzed (Participants) | 7 | 7
nM*hr
  Day 1 | 11701.0 (49.78) | 18953.4 (56.89)
  Day 14: number analyzed (Participants) | 7 | 4
  Day 14 | 20262.8 (71.34) | 30918.3 (55.68)
  Day 21: number analyzed (Participants) | 5 | 4
  Day 21 | 18264.9 (28.67) | 24515.6 (23.80)

20. Secondary Outcome: Terminal Half-Life (t1/2) for Alisertib 21 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Day 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Number analyzed (Participants) | 6 | 3
hr | 20.13 (6.326) | 26.13 (9.780)

21. Secondary Outcome: Accumulation Ratio (Rac) for Alisertib 21 Day Dosing
Description: Rac for Day 7=AUCt Day 7/AUCt Day 1. Rac for Day 14=AUCt Day 7/AUCt Day 1. Rac for Day 21=AUCt Day 21/AUCt Day 1.
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Days 14 and 21
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Number analyzed (Participants) | 7 | 7
ratio
  Day 14: number analyzed (Participants) | 7 | 4
  Day 14 | 2.482 (2.7166) | 2.103 (0.3861)
  Day 21: number analyzed (Participants) | 5 | 4
  Day 21 | 1.678 (0.7587) | 1.933 (1.1104)

22. Secondary Outcome: Peak/Trough Ratio for Aliserib 21 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Days 14 and 21
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Number analyzed (Participants) | 7 | 7
ratio
  Day 14: number analyzed (Participants) | 7 | 4
  Day 14 | 4.070 (2.4751) | 3.628 (0.4864)
  Day 21: number analyzed (Participants) | 5 | 4
  Day 21 | 4.792 (2.5652) | 4.658 (2.1825)

23. Secondary Outcome: CLss/F: Apparent Oral Clearance at Steady State 21 Day Dosing
Time Frame: Cycle 1: Pre-dose and multiple time-points (up to 10 hours) on Days 14 and 21
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Number analyzed (Participants) | 7 | 7
L/hr
  Day 14: number analyzed (Participants) | 7 | 4
  Day 14 | 4.753 (70.5636) | 4.364 (47.3164)
  Day 21: number analyzed (Participants) | 5 | 4
  Day 21 | 5.276 (28.1356) | 5.593 (21.8384)

24. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy Mitotic Index 7 Day Dosing
Description: Mitotic index was defined as the mean number of mitotic cells per millimeter (mm) length of the basoepithelial layer (BEL). Mitotic cells were counted manually within the BEL of 4, 5 micrometer (µm) skin sections stained with fluorescent-tagged antibodies specific to 2 mitotic markers; histone H3 phosphorylated on serine 10 (pHistH3) and MPM2. Deoxyribonucleic acid (DNA) was stained with a fluorescent marker as well. A positive change from Baseline indicates improvement.
Time Frame: Cycle 1: Pre-dose (Baseline) and Day 1, 6 hours post-dose; Day 7, 6 and 24 hours post-dose.
Population: Pharmacodynamics Evaluable Population was defined as all participants who received at least first dose of alisertib, had a baseline skin punch biopsy sample, and had at least 1 additional skin punch biopsy taken during Cycle 1 of treatment. Here number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: cells/mm
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D
Number analyzed (Participants) | 3 | 3 | 3 | 13 | 6 | 3 | 6
cells/mm
  Day 1, 6 Hours Post-Dose: number analyzed (Participants) | 3 | 3 | 3 | 13 | 6 | 2 | 6
  Day 1, 6 Hours Post-Dose | 0.187 (0.0709) | 0.107 (0.0777) | 0.197 (0.0814) | 0.310 (0.2087) | 0.378 (0.4107) | 0.175 (0.2333) | 0.850 (1.0741)
  Day 7, 6 Hours Post-Dose: number analyzed (Participants) | 3 | 3 | 3 | 11 | 6 | 3 | 6
  Day 7, 6 Hours Post-Dose | 0.193 (0.1650) | 0.617 (0.7514) | 2.703 (0.7112) | 3.489 (2.6893) | 6.220 (5.7549) | 8.757 (4.0493) | 9.150 (8.9050)
  Day 7, 24 Hours Post-Dose: number analyzed (Participants) | 3 | 3 | 2 | 9 | 1 | 2 | 3
  Day 7, 24 Hours Post-Dose | 0.140 (0.1179) | 0.397 (0.2159) | 5.270 (3.8325) | 3.184 (4.4984) | 1.250 (0.0000) | 25.190 (1.7678) | 17.123 (9.4877)

25. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy Mitotic Index 14 Day Dosing
Description: as for outcome 24
Time Frame: Cycle 1: Pre-dose (Baseline) and Day 1 and 7, 6 hours post-dose; Day 14, 6 and 24 hours post-dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: cells/mm
Arm/Group | Alisertib 50 mg QD 14D
Number analyzed (Participants) | 7
cells/mm
  Day 1, 6 Hours Post-Dose: number analyzed (Participants) | 1
  Day 1, 6 Hours Post-Dose | 1.180 (0.0000)
  Day 7, 6 Hours Post-Dose: number analyzed (Participants) | 5
  Day 7, 6 Hours Post-Dose | 0.950 (0.9963)
  Day 14, 6 Hours Post-Dose: number analyzed (Participants) | 5
  Day 14, 6 Hours Post-Dose | 1.146 (1.6239)
  Day 7, 24 Hours Post-Dose: number analyzed (Participants) | 4
  Day 7, 24 Hours Post-Dose | 0.368 (0.4464)

26. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy Mitotic Index 21 Day Dosing
Description: as for outcome 24
Time Frame: Cycle 1: Pre-dose (Baseline) and Day 7, 14 and 21, 6 hours post-dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: cells/mm
Arm/Group | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Number analyzed (Participants) | 7 | 7
cells/mm
  Day 7, 6 Hours Post-Dose | 1.534 (1.9201) | 1.900 (2.2774)
  Day 14, 6 Hours Post-Dose: number analyzed (Participants) | 7 | 5
  Day 14, 6 Hours Post-Dose | 0.341 (0.3182) | 1.168 (0.7587)
  Day 21, 6 Hours Post-Dose: number analyzed (Participants) | 5 | 4
  Day 21, 6 Hours Post-Dose | 0.250 (1.453) | 0.565 (0.5565)

27. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy Apoptotic Index 7 Day Dosing
Description: Apoptotic index was defined as the mean number of apoptotic cells per mm length of the basoepithelial layer (BEL). Apoptotic cells were counted manually within the BEL of 4, 5 µm skin sections stained with hematoxylin and eosin. A positive change from Baseline indicates improvement.
Time Frame: Cycle 1: Day 1, 6 hours post-dose; Days 7 6 and 24 hours post-dose; Day 21: 6 hours post-dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: cells/mm
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D
Number analyzed (Participants) | 3 | 3 | 3 | 13 | 6 | 3 | 6
cells/mm
  Day 1, 6 hour post-dose: number analyzed (Participants) | 3 | 3 | 3 | 13 | 6 | 2 | 6
  Day 1, 6 hour post-dose | 0.080 (0.0693) | 0.000 (0.0000) | 0.097 (0.0850) | 0.040 (0.0634) | 0.000 (0.0000) | 0.055 (0.0778) | 0.242 (0.2566)
  Day 7, 6 hour post-dose: number analyzed (Participants) | 3 | 3 | 3 | 11 | 6 | 3 | 6
  Day 7, 6 hour post-dose | 0.040 (0.0693) | 0.560 (0.9699) | 1.303 (0.5950) | 1.525 (2.2399) | 3.173 (4.3170) | 6.040 (1.9928) | 5.162 (2.2801)
  Day 7, 24 hour post-dose: number analyzed (Participants) | 3 | 3 | 2 | 9 | 1 | 2 | 3
  Day 7, 24 hour post-dose | 0.040 (0.0693) | 0.343 (0.4944) | 2.145 (1.6476) | 1.050 (1.749) | 0.830 (0.00) | 7.715 (0.1202) | 4.713 (1.1924)

28. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy Apoptotic Index 14 Day Dosing
Description: as for outcome 27
Time Frame: Cycle 1: Pre-dose (Baseline) and Day 1, 6 hours post-dose; Days 7 and 14, 6 and 24 hours post-dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: cells/mm
Arm/Group | Alisertib 50 mg QD 14D
Number analyzed (Participants) | 7
cells/mm
  Day 1, 6 hours post-dose: number analyzed (Participants) | 1
  Day 1, 6 hours post-dose | 0.000 (0.000)
  Day 7, 6 hours post-dose: number analyzed (Participants) | 5
  Day 7, 6 hours post-dose | 0.390 (0.8721)
  Day 14, 6 hours post-dose: number analyzed (Participants) | 5
  Day 14, 6 hours post-dose | 0.484 (0.7869)
  Day 14, 24 hours post-dose: number analyzed (Participants) | 4
  Day 14, 24 hours post-dose | 0.260 (0.3834)

29. Secondary Outcome: Change From Baseline in Alisertib Skin Punch Biopsy Apoptotic Index 21 Day Dosing
Description: as for outcome 27
Time Frame: Cycle 1: Pre-dose (Baseline) and Day 1, 6 hours post-dose; Days 7 and 14, 6 and 24 hours post-dose; Day 21: 6 hours post-dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: cells/mm
Arm/Group | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Number analyzed (Participants) | 7 | 7
cells/mm
  Day 7, 6 hours post-dose | 0.606 (0.9954) | 0.379 (0.6276)
  Day 14, 6 hours post-dose: number analyzed (Participants) | 7 | 5
  Day 14, 6 hours post-dose | 0.146 (0.2355) | 0.404 (0.4334)
  Day 21, 6 hours post-dose: number analyzed (Participants) | 5 | 4
  Day 21, 6 hours post-dose | 0.134 (0.1698) | 0.230 (0.1283)

30. Secondary Outcome: Change From Baseline in Alisertib Tumor Biopsy Mitotic Index 7 Day Dosing
Description: Tumor biopsy sections were immunoflourescently labeled with proliferative marker Ki67 and mitotic marker pHistH3. DNA was stained with a fluorescent marker as well. The Mitotic index was determined from the percentage of pHistH3 immunopositive cells within the Ki67 positive area. A positive change from Baseline indicates improvement.
Time Frame: Cycle 1: Pre-dose (Baseline) and Days 1 and 7, 6 hours post-dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D
Number analyzed (Participants) | 3 | 3 | 3 | 13 | 6 | 3 | 6
percentage of cells
  Day 1, 6 hours post-dose: number analyzed (Participants) | 2 | 1 | 2 | 5 | 2 | 1 | 3
  Day 1, 6 hours post-dose | 0.125 (0.1061) | 0.610 (0.0000) | 6.460 (9.1075) | 1.464 (1.3294) | 1.080 (0.3394) | 0.090 (0.0000) | 2.907 (2.0284)
  Day 7, 6 hours post-dose: number analyzed (Participants) | 2 | 1 | 2 | 5 | 2 | 1 | 3
  Day 7, 6 hours post-dose | 1.145 (0.0354) | 0.590 (0.0000) | 15.500 (13.5623) | 2.020 (2.9567) | 3.115 (3.1608) | 5.840 (0.0000) | 3.527 (2.1258)

31. Secondary Outcome: Change From Baseline in Alisertib Tumor Biopsy Mitotic Index 14 Day Dosing
Description: as for outcome 30
Time Frame: Cycle 1: Pre-dose (Baseline) and Day 7, 6 hours post-dose
Population: Pharmacodynamics Evaluable Population was defined as all participants who received at least the first dose of alisertib, had a baseline skin punch biopsy sample, and had at least 1 additional skin punch biopsy taken during Cycle 1 of treatment.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Alisertib 50 mg QD 14D
Number analyzed (Participants) | 7
percentage of cells | 0.008 (0.0000)

32. Secondary Outcome: Change From Baseline in Alisertib Tumor Biopsy Mitotic Index 21 Day Dosing
Description: as for outcome 30
Time Frame: Cycle 1: Pre-dose (Baseline) and Days 7 and 21, 6 hours post-dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Number analyzed (Participants) | 7 | 7
percentage of cells
  Day 7, 6 hours post-dose: number analyzed (Participants) | 3 | 4
  Day 7, 6 hours post-dose | 0.027 (0.0171) | 0.050 (0.0243)
  Day 21, 6 hours post-dose: number analyzed (Participants) | 2 | 2
  Day 21, 6 hours post-dose | 0.014 (0.0072) | 0.054 (0.0038)

33. Other Pre Specified Outcome: Percentage of Participants With Polymorphisms in Gene Encoding Enzyme UGT1A1
Description: A blood sample was collected prior to alisertib dosing for the purpose of genotyping for polymorphisms in UGT1A1. The percentage of participants in the polymorphism categories: wt/wt, wt/*28, *28/*28, *28/wt, *28/other and other/other is reported. wt=wild type. *28 polymorphism in the promoter region of a UGT1A1 allele resulting in reduced UGT1A1 expression.
Time Frame: Cycle 1: Pre-dose
Population: Safety population was defined as all participants who received any amount of study drug. A blood sample was not evaluable for 3 participants and was missing for 5 participants. Data is presented for one arm because the data was collected prior to the participant receiving their assigned treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib
Number analyzed (Participants) | 59
percentage of participants
  wt/wt | 34
  wt/*28 | 44
  *28/*28 | 7
  *28/wt | 0
  *28/other | 0
  other/other | 2

ADVERSE EVENTS:
Time Frame: Signing of the Informed Consent through 30 days following the last dose of study drug (up to 730 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alisertib 5 mg QD 7D | Alisertib 80 mg QD 7D | Alisertib 150 mg QD 7D | Alisertib 50 mg BID 7D | Alisertib 60 mg BID 7D | Alisertib 75 mg BID 7D | Alisertib 100 mg BID 7D | Alisertib 50 mg QD 14D | Alisertib 50 mg QD 21D | Alisertib 70 mg QD 21D
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/3 | 6/14 | 3/6 | 1/3 | 5/6 | 1/7 | 3/7 | 4/7
Other Adverse Events (participants affected / at risk) | 3/39 | 3/30 | 3/101 | 14/142 | 6/68 | 3/68 | 6/194 | 7/119 | 7/67 | 7/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alisertib 5 mg QD 7D (N=3) | Alisertib 80 mg QD 7D (N=3) | Alisertib 150 mg QD 7D (N=3) | Alisertib 50 mg BID 7D (N=14) | Alisertib 60 mg BID 7D (N=6) | Alisertib 75 mg BID 7D (N=3) | Alisertib 100 mg BID 7D (N=6) | Alisertib 50 mg QD 14D (N=7) | Alisertib 50 mg QD 21D (N=7) | Alisertib 70 mg QD 21D (N=7)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Alisertib 5 mg QD 7D (N=39) | Alisertib 80 mg QD 7D (N=30) | Alisertib 150 mg QD 7D (N=101) | Alisertib 50 mg BID 7D (N=142) | Alisertib 60 mg BID 7D (N=68) | Alisertib 75 mg BID 7D (N=68) | Alisertib 100 mg BID 7D (N=194) | Alisertib 50 mg QD 14D (N=119) | Alisertib 50 mg QD 21D (N=67) | Alisertib 70 mg QD 21D (N=68)
Nausea (Gastrointestinal disorders) | 1/3 (3) | 0/3 (0) | 2/3 (8) | 1/14 (1) | 2/6 (2) | 1/3 (1) | 4/6 (9) | 2/7 (2) | 3/7 (6) | 5/7 (5)
Stomatitis (Gastrointestinal disorders) | 0/3 (0) | 1/3 (1) | 2/3 (6) | 3/14 (3) | 2/6 (2) | 2/3 (7) | 3/6 (6) | 0/7 (0) | 3/7 (3) | 1/7 (1)
Diarrhoea (Gastrointestinal disorders) | 1/3 (4) | 0/3 (0) | 1/3 (2) | 2/14 (2) | 3/6 (3) | 2/3 (4) | 2/6 (9) | 1/7 (3) | 2/7 (4) | 2/7 (3)
Vomiting (Gastrointestinal disorders) | 1/3 (5) | 0/3 (0) | 1/3 (4) | 0/14 (0) | 2/6 (3) | 1/3 (1) | 3/6 (3) | 3/7 (4) | 2/7 (7) | 3/7 (3)
Abdominal pain (Gastrointestinal disorders) | 0/3 (0) | 1/3 (1) | 1/3 (1) | 1/14 (2) | 2/6 (2) | 0/3 (0) | 2/6 (3) | 3/7 (3) | 0/7 (0) | 0/7 (0)
Dyspepsia (Gastrointestinal disorders) | 1/3 (1) | 0/3 (0) | 1/3 (2) | 0/14 (0) | 1/6 (1) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 1/7 (1) | 1/7 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2/3 (2) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 1/6 (3) | 0/3 (0) | 0/6 (0) | 2/7 (2) | 0/7 (0) | 0/7 (0)
Constipation (Gastrointestinal disorders) | 1/3 (1) | 0/3 (0) | 1/3 (2) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 3/7 (3)
Enteritis (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 3/14 (3) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 2/7 (4) | 0/7 (0) | 0/7 (0)
Dry mouth (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 2/6 (2) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Proctalgia (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 1/3 (1) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 3/6 (4) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 1/3 (2) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 2/6 (5) | 0/7 (0) | 0/7 (0) | 1/7 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 1/3 (1) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 2/6 (3) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Anal fissure (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 2/6 (2) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Haematochezia (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Abdominal distension (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Ascites (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Colonic haemorrhage (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Dysphagia (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Flatulence (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 1/6 (1) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Haemorrhoids (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Odynophagia (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Oral pain (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Perianal erythema (Gastrointestinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Anaemia (Blood and lymphatic system disorders) | 2/3 (2) | 2/3 (3) | 2/3 (3) | 8/14 (11) | 4/6 (4) | 3/3 (4) | 5/6 (6) | 5/7 (6) | 4/7 (4) | 1/7 (1)
Leukopenia (Blood and lymphatic system disorders) | 0/3 (0) | 1/3 (2) | 2/3 (8) | 8/14 (11) | 3/6 (3) | 2/3 (7) | 6/6 (9) | 2/7 (3) | 1/7 (1) | 4/7 (4)
Neutropenia (Blood and lymphatic system disorders) | 0/3 (0) | 1/3 (1) | 3/3 (9) | 4/14 (5) | 4/6 (6) | 2/3 (7) | 3/6 (8) | 2/7 (2) | 3/7 (4) | 2/7 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0/3 (0) | 0/3 (0) | 2/3 (4) | 9/14 (11) | 2/6 (2) | 1/3 (1) | 0/6 (0) | 6/7 (10) | 2/7 (2) | 0/7 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0/3 (0) | 1/3 (1) | 2/3 (5) | 5/14 (8) | 2/6 (4) | 1/3 (3) | 5/6 (6) | 2/7 (4) | 0/7 (0) | 1/7 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0/3 (0) | 0/3 (0) | 1/3 (3) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Anorexia (Metabolism and nutrition disorders) | 2/3 (2) | 0/3 (0) | 2/3 (5) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 2/6 (8) | 1/7 (1) | 4/7 (4) | 2/7 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0/3 (0) | 1/3 (1) | 0/3 (0) | 3/14 (4) | 1/6 (1) | 0/3 (0) | 2/6 (2) | 2/7 (4) | 0/7 (0) | 1/7 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 5/14 (5) | 1/6 (1) | 0/3 (0) | 0/6 (0) | 2/7 (2) | 0/7 (0) | 0/7 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0/3 (0) | 1/3 (1) | 0/3 (0) | 3/14 (6) | 1/6 (1) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 1/7 (1) | 1/7 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1/3 (1) | 0/3 (0) | 0/3 (0) | 3/14 (3) | 2/6 (2) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0/3 (0) | 1/3 (2) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 3/7 (5) | 0/7 (0) | 0/7 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1/3 (1) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 2/6 (2) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Hyperproteinaemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 2/7 (2) | 0/7 (0) | 0/7 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 2/14 (4) | 1/6 (1) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 2/14 (3) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 1/3 (1) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Hyperchloraemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 2/7 (3) | 0/7 (0) | 0/7 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 2/14 (2) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 2/6 (2) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Dehydration (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Fluid intake reduced (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Blood alkaline phosphatase increased (Investigations) | 1/3 (1) | 1/3 (1) | 0/3 (0) | 5/14 (6) | 0/6 (0) | 1/3 (1) | 4/6 (4) | 3/7 (3) | 0/7 (0) | 2/7 (2)
Alanine aminotransferase increased (Investigations) | 0/3 (0) | 1/3 (1) | 0/3 (0) | 7/14 (8) | 1/6 (1) | 1/3 (1) | 1/6 (1) | 3/7 (5) | 1/7 (1) | 1/7 (1)
Aspartate aminotransferase increased (Investigations) | 1/3 (1) | 0/3 (0) | 0/3 (0) | 4/14 (6) | 2/6 (2) | 0/3 (0) | 0/6 (0) | 2/7 (3) | 1/7 (1) | 2/7 (2)
Gamma-glutamyltransferase increased (Investigations) | 0/3 (0) | 1/3 (1) | 0/3 (0) | 4/14 (4) | 0/6 (0) | 1/3 (1) | 3/6 (3) | 2/7 (3) | 0/7 (0) | 1/7 (1)
Blood creatinine increased (Investigations) | 1/3 (1) | 0/3 (0) | 0/3 (0) | 2/14 (2) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 1/7 (1) | 0/7 (0) | 1/7 (1)
Blood bilirubin increased (Investigations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 1/3 (1) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Blood urea increased (Investigations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 2/14 (2) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Platelet count decreased (Investigations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 1/7 (1) | 0/7 (0)
Blood creatinine decreased (Investigations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Red blood cell count decreased (Investigations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Transaminases increased (Investigations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 1/3 (1) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Weight decreased (Investigations) | 1/3 (1) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Asthenia (General disorders) | 3/3 (3) | 0/3 (0) | 2/3 (9) | 3/14 (3) | 3/6 (3) | 2/3 (2) | 5/6 (10) | 3/7 (3) | 6/7 (6) | 4/7 (4)
Pyrexia (General disorders) | 0/3 (0) | 0/3 (0) | 1/3 (4) | 1/14 (1) | 1/6 (1) | 1/3 (1) | 5/6 (8) | 4/7 (5) | 1/7 (1) | 2/7 (2)
Oedema peripheral (General disorders) | 1/3 (1) | 0/3 (0) | 1/3 (1) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 1/7 (1)
Chills (General disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 2/6 (2) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Chest pain (General disorders) | 1/3 (1) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 1/7 (1)
Feeling jittery (General disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Gait disturbance (General disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Red man syndrome (General disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Somnolence (Nervous system disorders) | 1/3 (1) | 2/3 (2) | 2/3 (8) | 4/14 (4) | 2/6 (3) | 1/3 (6) | 3/6 (10) | 0/7 (0) | 1/7 (1) | 5/7 (5)
Headache (Nervous system disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 1/7 (1) | 1/7 (1) | 2/7 (2)
Cerebral ataxia (Nervous system disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 2/7 (2)
Dizziness (Nervous system disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 1/6 (2) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Aphonia (Nervous system disorders) | 0/3 (0) | 1/3 (1) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Dysaesthesia (Nervous system disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 1/6 (1) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Dysgeusia (Nervous system disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 1/6 (1) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Neuropathic pain (Nervous system disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 1/6 (1) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Paraesthesia (Nervous system disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 1/7 (1) | 0/7 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0/3 (0) | 2/3 (2) | 3/3 (3) | 1/14 (1) | 4/6 (4) | 2/3 (2) | 4/6 (4) | 1/7 (1) | 3/7 (3) | 5/7 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 2/6 (2) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 1/6 (1) | 1/3 (2) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 1/3 (1) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Rash (Skin and subcutaneous tissue disorders) | 1/3 (1) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Blister (Skin and subcutaneous tissue disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0/3 (0) | 0/3 (0) | 1/3 (1) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0/3 (0) | 0/3 (0) | 1/3 (1) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Nasopharyngitis (Infections and infestations) | 1/3 (1) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 1/6 (1) | 2/3 (2) | 3/6 (3) | 2/7 (2) | 1/7 (2) | 0/7 (0)
Oral candidiasis (Infections and infestations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 1/3 (1) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Respiratory tract infection (Infections and infestations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 1/7 (2) | 0/7 (0)
Bronchitis (Infections and infestations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Catheter related infection (Infections and infestations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Gastroenteritis escherichia coli (Infections and infestations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Herpes simplex (Infections and infestations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 1/7 (1)
Nail infection (Infections and infestations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Urinary tract infection (Infections and infestations) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/3 (1) | 1/3 (1) | 1/3 (1) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 1/7 (1) | 1/7 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0/3 (0) | 2/3 (2) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 2/7 (2) | 0/7 (0) | 0/7 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/3 (0) | 0/3 (0) | 1/3 (1) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 1/7 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0/3 (0) | 1/3 (1) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 1/7 (2) | 0/7 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/3 (0) | 0/3 (0) | 1/3 (1) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0/3 (0) | 1/3 (1) | 1/3 (1) | 0/14 (0) | 1/6 (1) | 0/3 (0) | 0/6 (0) | 2/7 (2) | 1/7 (1) | 1/7 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (2) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0/3 (0) | 1/3 (1) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/3 (0) | 0/3 (0) | 1/3 (1) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1/3 (1) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Insomnia (Psychiatric disorders) | 0/3 (0) | 0/3 (0) | 1/3 (1) | 0/14 (0) | 1/6 (1) | 2/3 (4) | 3/6 (4) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Confusional state (Psychiatric disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 2/6 (2) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Affect lability (Psychiatric disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Anxiety (Psychiatric disorders) | 0/3 (0) | 0/3 (0) | 1/3 (1) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Bradyphrenia (Psychiatric disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 1/7 (1)
Nervousness (Psychiatric disorders) | 1/3 (1) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Keratitis (Eye disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 1/6 (1) | 2/3 (3) | 2/6 (12) | 0/7 (0) | 1/7 (1) | 0/7 (0)
Dry eye (Eye disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 1/6 (1) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Vision blurred (Eye disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3 (2) | 0/3 (0) | 0/3 (0) | 1/14 (1) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 2/7 (2) | 0/7 (0)
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 1/7 (1) | 0/7 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 1/3 (3) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Hepatic pain (Hepatobiliary disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 2/14 (2) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0/3 (0) | 1/3 (2) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 1/7 (2)
Jaundice (Hepatobiliary disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 1/3 (1) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Haematuria (Renal and urinary disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 1/7 (1) | 0/7 (0)
Dysuria (Renal and urinary disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Oliguria (Renal and urinary disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Pollakiuria (Renal and urinary disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 1/7 (1)
Hypotension (Vascular disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Haematoma (Vascular disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 1/6 (1) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Phlebitis (Vascular disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 1/7 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 1/7 (1) | 0/7 (0)
Palpitations (Cardiac disorders) | 0/3 (0) | 1/3 (1) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 0/7 (0) | 0/7 (0) | 0/7 (0)
Ear pain (Ear and labyrinth disorders) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/14 (0) | 0/6 (0) | 0/3 (0) | 0/6 (0) | 1/7 (1) | 0/7 (0) | 0/7 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.